CLINICAL TRIAL: NCT00991536
Title: Impact of Non Invasive Ventilation on Quality of Sleep
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Rodenstein D. / Professor, Cliniques Universitaires Saint-Luc
Other Study IDs: B40320084384
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Restrictive Pulmonary Disorders; Non Invasive Ventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic respiratory failure: Patients with restrictive pulmonary disorders leading to progressive hypercapnic respiratory failure and requiring nocturnal non-invasive ventilation

SUMMARY:
Quality of sleep is profoundly affected in patients with hypercapnic respiratory failure and restrictive disorders, with a decrease in rapid eye movement (REM) and slow wave sleep, and an increase in sleep fragmentation. Assisted ventilation aims at improving blood gases, but may also have a favorable impact on sleep structure. The investigators reviewed polysomnographic and blood gas data obtained between 1987 and 2008 in 95 patients with restrictive pulmonary disorders, before and after implementing non-invasive ventilatory support.

DETAILED DESCRIPTION:
Chart review of all patients with predominantly restrictive pulmonary disorders treated for respiratory failure by NIV at our institution between 1987 and 2008.

Data systematically recorded included pulmonary function tests, diurnal arterial blood gases, and polysomnography before and after implementation of nocturnal NIV.

ELIGIBILITY:
Inclusion Criteria:

* Patients with restrictive pulmonary disorders (neuro-muscular diseases, chest wall disorders, sequellae of tuberculosis) leading to hypercapnic respiratory failure requiring non invasive ventilation (NIV), investigated according to clinical standards in our institution by polysomnography before and after implementation of NIV

Exclusion Criteria:

* Patients fulfilling inclusion criteria for whom diagnostic polysomnography and/or polysomnography under NIV were not performed

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with respiratory failure due to predominantly restrictive disorders submitted to NIV in preparation for long-term home ventilation and assessed between 1987 and 2008 at the Sleep laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 1987-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Daytime arterial blood gases and Polysomnography before and after non invasive ventilation | Average of 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rodenstein, Professor, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain